CLINICAL TRIAL: NCT06231966
Title: Randomized Comparison of Efficacy and Safety of High-intensity Rosuvastatin/Ezetimibe Combination Versus Treat-to-target Rosuvastatin Monotherapy for Patients With Peripheral Artery or Polyvascular Disease (CARE-PVD Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1212
Record Dates: First submitted 2023-12-08; First posted 2024-01-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Artery Disease; Polyvascular Disease
Keywords: Peripheral artery disease; polyvascular disease; lipid lowering therapy; LDL cholesterol; Clinical outcomes
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin/ezetimibe combination therapy (Experimental): Combination therapy of high-intensity dose rosuvastatin and ezetimibe
  Interventions: Drug: Combination therapy of high-intensity dose rosuvastatin and ezetimibe
- Rosuvastatin monotherapy (Active Comparator): Rosuvastatin monotherapy for treat-to-target (LDL cholesterol < 70 mg/dL)
  Interventions: Drug: Rosuvastatin monotherapy for treat-to-target

INTERVENTIONS:
Drug: Combination therapy of high-intensity dose rosuvastatin and ezetimibe — Combination therapy of rosuvastatin 20 mg and ezetimibe 10 mg
  Arms: Rosuvastatin/ezetimibe combination therapy
Drug: Rosuvastatin monotherapy for treat-to-target — Rosuvastatin monotherapy for treat-to-target (LDL cholesterol <70 mg/dL)
  Arms: Rosuvastatin monotherapy

SUMMARY:
Patients with atherosclerotic peripheral artery disease often have combined coronary artery disease or cerebral artery disease and show high rates of cardiovascular mortality and morbidities. Therefore, secondary prevention for these patients is of great clinical importance. Currently, Korean, US, and European guidelines recommend different LDL cholesterol target goals in patients with peripheral artery disease. In recent clinical trials, combination therapy of statin plus ezetimibe demonstrated improved cardiovascular outcomes compared with statin monotherapy. Thus, the purpose of the CARE-PVD study is to investigate whether the combination therapy of high intensity rosuvastatin 20 mg plus ezetimibe 10 mg can improve cardiovascular outcomes in patient with peripheral artery disease or polyvascular artery disease in comparison with rosuvastatin treat-to-target (LDL cholesterol <70 mg/dL) monotherapy.

DETAILED DESCRIPTION:
* A multicenter prospective randomized controlled clinical trial
* A total of 2462 subjects with cperipheral artery disease or polyvascular disease will be included according to inclusion and exclusion criteria.
* Patients will be randomized in a 1:1 manner into the rosuvastatin/ezetimibe combination therapy group or rosuvastatin monotherapy group. • The randomization will be startified by previous use of statin and presence of diabetes mellitus. • In the rosuvastatin/ezetimibe combination therapy group, rosuvastatin 20 mg plus ezetimibe 10 mg will be administered. • In the rosuvastatin monotherapy group, rosuvastatin will be administered and the dose of rosuvastatin will be adjusted to attain the target LDL cholesterol level < 70 mg/dL.
* Patients will be followed clinically for 3years.
* The primary endpoint is defined as the composite of Major cardiovascular event (MACE) or major adverse limb event (MALE) at 3-year follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Ages 19-80
2. Patient with arteriosclerotic lower extremity artery disease or multivessel disease 1) Arteriosclerotic lower extremity artery disease: If any of the following applies

   * Ankle-brachial index <0.85 with symptoms of intermittent claudication
   * Lower extremity artery stenosis of more than 50% on imaging tests
   * History of receiving interventional or surgical treatment for lower extremity artery disease) 2) Arteriosclerotic multivessel disease: When at least two of the following diseases exist even if there is no lower extremity artery disease
   * Coronary artery disease
   * History of carotid artery stenosis (more than 50%) or ischemic stroke/transient cerebral ischemia event
   * degenerative thoracic (maximum diameter >4 cm) or abdominal (maximum diameter >3cm) aortic aneurysm
3. Patients on medication for dyslipidemia or patients with LDL cholesterol level higher than the target level for peripheral arterial disease (≥70 mg/dL) and not on lipid lowering medication

Exclusion criteria:

1. Chronic limb threatening ischemia (Rutherford 4~6)
2. History of acute coronary syndrome or stroke/TIA or lower extremity amputation within 6 months
3. Acute liver disease or persistent unexplained elevation of serum AST or ALT more than twice the upper limit of normal
4. Severe renal dysfunction (eGFR <30 mL/min/1.73m2) or dependancy on dialysis
5. History of allergic or hypersensitivity reaction to statin or ezetimibe or side effects requiring discontinuation of lipid lowering therapy
6. Solid organ transplant recipients
7. Pregnant women, potentially pregnant or lactating women
8. Life expectancy of less than 3 years
9. When follow-up for more than 1 year is not possible
10. Inability to understand or read the consent form

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2462 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2029-05-06 (Estimated)

PRIMARY OUTCOMES:
Composite of Major cardiovascular event or major adverse limb event | at 3 years
  Composite of Major cardiovascular event (MACE) or major adverse limb event (MALE) at 3-year follow-up MACE includes death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, coronary revascularization, and hospitalization for unstable angina or heart failure. MALE includes acute lower extremity ischemia, major lower extremity amputation, and revascularization of lower extremity arteries.

SECONDARY OUTCOMES:
Major cardiovascular event(death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, coronary revascularization, and hospitalization for unstable angina or heart failure) | at 1, 2, and 3 years
  Major cardiovascular event(death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, coronary revascularization, and hospitalization for unstable angina or heart failure)
Major adverse limb event(acute lower extremity ischemia, major lower extremity amputation, and revascularization of lower extremity arteries) | at 1, 2, and 3 years
  Major adverse limb event(acute lower extremity ischemia, major lower extremity amputation, and revascularization of lower extremity arteries)
discontinuation of lipid lowering therapy | at 1, 2, and 3 years
  Intolerance of lipid lowering therapy
adverse clinical events related to lipid lowering therapy | at 1, 2, and 3 years
  adverse clinical events related to lipid lowering therapy
attainment of LDL cholesterol | at 1, 2, and 3 years
  attainment of LDL cholesterol goal
Major cardiovascular event : non-fatal myocardial infarction | at 1, 2, and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No